CLINICAL TRIAL: NCT07170124
Title: The Effect of Obstetric Exercises on Depression, Pregnancy Complaints and Quality of Life: A Randomized Controlled Trial
Brief Title: Obstetric Exercise and Maternal Outcomes in Pregnancy
Acronym: BDI-PSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Asst. Prof., Bingol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-33117789-044-126827
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Depression During Pregnancy; Pregnancy; Pregnancy Complications
Keywords: Obstetric exercise; Depression; Pregnancy symptoms; Quality of life
MeSH Terms: conditions — Pregnancy Complications; Depression

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants in the intervention group will take part in a four-week obstetric exercise program designed specifically for pregnant women. The program will be led by a licensed physiotherapist and delivered in small group sessions at the hospital's pregnancy school. Exercises will focus on relaxation, breathing techniques, stretching, posture correction, and low-impact strengthening movements appropriate for pregnancy. Sessions will be closely supervised to ensure safety and adapted to each participant's gestational stage and physical capacity. In addition to routine prenatal care, participants in this group will receive structured, physiotherapist-led exercise sessions once a week for four weeks.
  Interventions: Other: Obstetric exercises
- Control group (No Intervention): Participants in the control group will receive routine prenatal care provided by the hospital's antenatal clinic and pregnancy school. This includes standard obstetric follow-up, regular health check-ups, and educational counseling typically offered during pregnancy, but no structured obstetric exercise program.

INTERVENTIONS:
Other: Obstetric exercises — The intervention will consist of a structured obstetric exercise program administered by a physiotherapist who is permanently employed at the hospital's prenatal education center, ensuring the reliability and standardization of the intervention. The program will be based on the "Pregnancy and Exercise Guide" (2012) published by the Turkish Ministry of Health and will be delivered in the pregnancy school of a public hospital in eastern Türkiye.
  The exercises will be provided at weekly intervals and will include:
  Active joint movements to improve mobility and maintain functional range of motion,
  Stretching exercises to enhance flexibility and alleviate musculoskeletal discomfort,
  Calisthenic bodyweight exercises to promote muscle strength and endurance,
  Relaxation and breathing techniques to reduce stress and improve maternal well-being.
  Arms: Exercise group

SUMMARY:
This randomized controlled trial will be conducted in the antenatal clinic and pregnancy school of a public hospital in eastern Türkiye. The study will aim to investigate the effects of obstetric exercises on depression, pregnancy-related complaints, and quality of life in women receiving prenatal care.

A total of 100 pregnant women will be recruited and randomly assigned to either the intervention group (n=50) or the control group (n=50). The intervention group will participate in a four-week, physiotherapist-led, closely supervised obstetric exercise program, while the control group will continue to receive routine prenatal care.

Data will be collected through a sociodemographic questionnaire, the Beck Depression Inventory (BDI), and the Pregnancy Symptoms Inventory (PSI). Post-intervention outcomes will be analyzed using independent-samples t-tests to compare groups, and multiple linear regression will be applied to determine the influence of sociodemographic factors on study variables.

This study is expected to contribute to the evidence base by clarifying the potential role of obstetric exercise in reducing depressive symptoms, alleviating pregnancy complaints, and improving maternal quality of life within routine prenatal care settings.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate the effectiveness of a structured obstetric exercise program on maternal mental health and pregnancy-related outcomes. The study will be conducted in the antenatal clinic and pregnancy school of a public hospital in eastern Türkiye, with a total of 100 pregnant women enrolled. Participants will be randomly allocated into two parallel groups: an intervention group (n=50) and a control group (n=50). Randomization will be performed using a computer-generated allocation sequence to minimize selection bias.

The intervention consists of a four-week exercise program developed specifically for pregnant women, led and closely supervised by a physiotherapist trained in maternal health. Sessions will take place three times per week, each lasting approximately 45-60 minutes, and will include a combination of breathing exercises, stretching, posture training, and low-intensity strengthening movements adapted for pregnancy. Exercise intensity and duration will be progressively adjusted according to gestational age, maternal comfort, and current obstetric guidelines. To ensure safety, maternal vital signs and fetal well-being will be monitored before and after each session. Participants will also receive verbal instructions on safe daily activity modifications and home practice recommendations.

The control group will receive standard prenatal care provided by the antenatal clinic, without additional structured exercise training. Both groups will continue to have access to routine obstetric monitoring, counseling, and educational materials typically offered by the hospital's pregnancy school.

Primary data will be collected using validated self-report instruments:

Beck Depression Inventory (BDI): to assess depressive symptoms. Pregnancy Symptoms Inventory (PSI): to evaluate frequency and severity of common pregnancy-related complaints.

Sociodemographic Questionnaire: to capture baseline characteristics such as age, education, employment, and income.

Outcome assessments will be conducted at baseline (prior to randomization) and immediately after completion of the four-week program. Data analysis will include independent-samples t-tests to assess between-group differences in outcome measures. Multiple linear regression models will be applied to determine the potential influence of sociodemographic and clinical variables on depressive symptoms, pregnancy complaints, and quality of life scores. Statistical significance will be set at p<0.05.

Ethical approval has been obtained from the relevant institutional review board, and written informed consent will be secured from all participants prior to enrollment. All procedures will comply with the principles of the Declaration of Helsinki.

This study aims to provide more robust evidence on the contribution of physiotherapist-led obstetric exercise programs to maternal health. By focusing on depression, pregnancy-related complaints, and quality of life, the results are expected to inform clinical practice guidelines and support the integration of safe exercise interventions into routine prenatal care in Türkiye and similar healthcare contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Low-risk singleton pregnancy confirmed by ultrasound
* No chronic illness
* No psychiatric disorder
* No physical disability
* Voluntary agreement to participate in the study
* Gestational age between 28 and 42 weeks (third trimester)

Exclusion Criteria:

* Body mass index (BMI) ≥ 40 kg/m² or ≤ 18 kg/m²
* Concurrent participation in another exercise or psychosocial intervention study
* Failure to attend at least one exercise session

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Depression Symptoms Assessed by BDI | At enrollment
  The Beck Depression Inventory (BDI) is a 21-item self-report scale measuring depressive symptoms. Each item is scored from 0 to 3, yielding a total score ranging from 0 to 63. Higher scores indicate more severe depressive symptoms (0-13 minimal, 14-19 mild, 20-28 moderate, 29-63 severe). The mean change in BDI total score from baseline to post-intervention will be compared between groups.
Change in Pregnancy-Related Complaints Assessed by PSI | At enrollment
  Pregnancy Symptoms Inventory (PSI): The scale consists of 42 items assessing the frequency of symptoms commonly experienced during pregnancy (e.g., fatigue, nausea, vomiting, reflux, constipation, dry mouth, cravings, insomnia). Each item is rated for frequency (0=never to 3=often) and limitation (0=not at all to 3=quite a lot). Higher scores indicate greater frequency and severity of complaints. The mean change in PSI total score from baseline to post-intervention will be compared between groups.

SECONDARY OUTCOMES:
Change in Depression Symptoms Assessed by BDI | At baseline and immediately post-intervention (4 weeks)
  The Beck Depression Inventory (BDI) is a 21-item self-report scale measuring depressive symptoms. Each item is scored from 0 to 3, yielding a total score ranging from 0 to 63. Higher scores indicate more severe depressive symptoms (0-13 minimal, 14-19 mild, 20-28 moderate, 29-63 severe). The mean change in BDI total score from baseline to post-intervention will be compared between groups.
Change in Pregnancy-Related Complaints Assessed by PSI | At baseline and immediately post-intervention (4 weeks)
  Pregnancy Symptoms Inventory (PSI): The scale consists of 42 items assessing the frequency of symptoms commonly experienced during pregnancy (e.g., fatigue, nausea, vomiting, reflux, constipation, dry mouth, cravings, insomnia). Each item is rated for frequency (0=never to 3=often) and limitation (0=not at all to 3=quite a lot). Higher scores indicate greater frequency and severity of complaints. The mean change in PSI total score from baseline to post-intervention will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, Ph.D., Principal Investigator — Bingol University; Mesut Çelik, Ph.D., Study Director — Bingol University; Gülcan Çelik, Bachelor's Degree, Study Chair — Bingöl State Hospital
Locations (1):
- Bingöl State Hospital, Bingöl, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No